CLINICAL TRIAL: NCT03057990
Title: A Phase 1 Study of Pyrimethamine, a STAT3 Inhibitor, for the Treatment of Intermediate/ High-risk Myelodysplastic Syndromes (MDS) That Has Relapsed or is Refractory to Azanucleosides
Brief Title: Pyrimethamine for Intermediate/High-risk Myelodysplastic Syndromes (MDS)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never opened; closed on 06/29/2021 due to no enrllment
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10346
Record Dates: First submitted 2016-11-30; First posted 2017-02-20 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Pyrimethamine; Myelodysplastic Syndromes (MDS); Refractory; Relapsed
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pyrimethamine Treatment (Intra-patient) (Experimental): 50mg/100mg/150mg once daily on days 1-28 of each 28-day cycle. Administered using intra-patient dose escalation, starting at 50 mg and up to 150 mg.
  Interventions: Drug: Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine — Pyrimethamine will be administered 50mg/100mg/150mg once daily on days 1-28 of each 28-day cycle. Administered using intra-patient dose escalation, starting at 50 mg and up to 150 mg.
  Other Names: Daraprim

SUMMARY:
This is a phase I study designed to assess the maximum tolerated dose (MTD) of pyrimethamine and provide the recommended Phase 2 dose (RP2D) for the treatment of intermediate/high-risk MDS that is refractory to or relapsed after treatment with azanucleosides.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety, dose tolerance, pharmacokinetics and pharmacodynamics of pyrimethamine in intermediate / high-risk / relapsed or azanucleoside-refractory MDS within the confines of a phase I study.

Pyrimethamine self-administered by participants orally once per day in morning with food. Phase 1 study will start at dose of 50 mg once per day. (NOTE: For participants at dose level of 50mg, the dose reduction, if needed is 25 mg.)

Intra-patient dose escalation is permitted (not beyond the highest dose allowed) if Complete Remission/Response (CR) is not reached in week 1 of Cycle 3 and there is no significant toxicity. (NOTE: In this study, the term "intra-patient" indicates within each participant and not between different participants; i.e., dose escalation will be done within each individual participant.) The decision to escalate intra-patient doses will be based on safety and dose tolerance assessments made at the end of one treatment cycle (28 days of continuous drug administration) for all 6 participants. Dose-limiting toxicity (DLT) is defined as the occurrence of two consecutive grade 2 or 3 serious adverse events (SAEs) not recovered within 24 hours at a given dose. MTD will be defined as the dose where no DLT is observed among three consecutive participants, or no more than one DLT among six participants. Participants will be treated initially for one 28-day cycle followed by a toxicity evaluation - Toxicity and adverse effect assessments will be made on Day 1 and Day 28 of every cycle of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants at or above the age of 18 years
* Diagnosis of MDS confirmed within 6 months, by review of patient chart, prior to study entry according to WHO (World Health Organization) criteria or FAB (French-American-British) classification
* MDS classified as intermediate-1, intermediate-2 or high risk as per the International Prognostic Scoring System-Revised (IPSS-R) score with a confirmed diagnosis of MDS with cytogenetic abnormalities at diagnosis and bone marrow blast percentage between 10 and 30 percent (for patients with cytogenetic failure or dry tap)
* Potential participants must meet ONE of the following:

  * Progression (according to 2006 International Working Group (IWG) criteria) at any time after initiation of azacitidine or decitabine treatment during the past 3 years; OR
  * Failure to achieve complete or partial response or hematological improvement (according to 2006 IWG) after at least four cycles of azacitidine or decitabine administered during the past 3 years OR
  * Relapse after initial complete or partial response or hematological improvement (according to 2006 IWG criteria) observed after at least four cycles of azacitidine or decitabine administered during the past 3 years OR
  * Intolerance to azacitidine or decitabine defined by drug-related more than or equal to Grade 3 liver or renal toxicity leading to treatment discontinuation during the past 3 years
* Off all other treatments for MDS for at least 3 weeks. Filgrastim (G-CSF) and erythropoietin are allowed before and during the study as clinically indicated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Patient (or patient's legally authorized representative) must signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study
* Adequate organ and marrow function as defined in the protocol.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria:

* Current or anticipated use of other investigational agents
* Participants who have had chemotherapy or radiotherapy within 3 weeks prior to entering the study or those who have not recovered from clinically significant adverse events due to agents administered more than 3 weeks earlier.
* History of allergic reactions or sensitivity to pyrimethamine
* Patients with a history of folic acid deficiency, currently on folic acid replacement therapy or a previous history of megaloblastic anemia thought related to folic acid deficiency
* Current use or anticipated need for treatment with any medications or substances that are inhibitors or inducers of CYP2C9.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Day 28
  Determination of DLT to be made at the completion of each cohort.
Maximum tolerated dose (MTD) | up to 28 days
  The dose where no DLT is observed among 3 consecutive participants, or no more than one DLT among 6 participants.
Recommended Phase II Dose (RPTD, RP2D) | 12 months
  Pyrimethamine will be dose-escalated until the largest dose is reached that is determined to be safe based on adverse event reporting and dose-limiting toxicity information from all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Shastri, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No